CLINICAL TRIAL: NCT06025136
Title: The Effect of the Use of Gel Pillows on the Sleep Quality and General Comfort Levels of the Patients in the Preoperative Period
Brief Title: The Effect of the Use of Gel Pillows on the Sleep Quality and General Comfort Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Associate Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-PO198
Record Dates: First submitted 2023-01-24; First posted 2023-09-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Preoperative; Sleep; Comfort
Keywords: comfort; gel pillows; sleep quality; nursing care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The research will be conducted using randomized controlled, experimental type and single-blind research methods. For this purpose, after the data are collected, they will be coded as A and B groups, so the researcher who will make the research statistics will analyze the data without knowing the study and control groups. Randomization method will be used to determine the groups. For this, the patients who meet the study criteria and volunteer will be assigned to the groups using the randomization program 'Random Allocation Software 2.0' according to the order of hospitalization.
Who Masked: Outcomes Assessor
Masking Description: The data analyse is going to be completed by a independent researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who are visited in their rooms on the evening of the day before the surgery will be given a gel pillow with a cooling surface feature for night use. Patients will be asked to note the time they go to bed for a night's sleep and the time they wake up on the morning of the surgery. If patients stop using pillows at night, they will be asked to inform the investigator when they come to their room in the morning.Patients will be visited again on the morning of the surgery day.The Richard Campbell Sleep Scale was used to evaluate the nighttime sleep quality of the patients;General Comfort Scale to evaluate comfort.
  Interventions: Other: Using a gel pillow
- Control Group (No Intervention): The patients who were visited in their rooms on the evening of the day before the operation will be given pillows that have the same characteristics as the pillows that the patients in the study group will use, but do not have a gel surface, to use at night. Patients will be asked to note the time they go to bed for a night's sleep and the time they wake up on the morning of the surgery.Participants in the control group will receive no other interventions.Patients will be visited again on the morning of the surgery day.The Richard Campbell Sleep Scale was used to evaluate the nighttime sleep quality of the patients;General Comfort Scale to evaluate comfort levels.

INTERVENTIONS:
Other: Using a gel pillow — Within the scope of the study, gel pillows with a cold surface were used in the patients in the study group. It is produced by combining the obtained special liquid with elastic material with NASA approved molecule exchange technology and is made of OEKO-TEX CLASS 1 certified material.Thanks to the gel material on the pillow surface, the surface temperature is reduced from 37°C to 24°C in about 10 seconds. It gives a feeling of coolness with its thermal conductivity feature.
  Arms: Intervention Group

SUMMARY:
The study was conducted to evaluate the effect of using gel pillows on the sleep quality and general comfort levels of patients in the preoperative period.The main hypotheses are:

H1: 'The sleep quality of patients who use gel pillows in the preoperative period is higher than those who do not use gel pillows' H2: "The general comfort level of the patients who used gel pillows in the preoperative period is higher than those who did not use gel pillows".

Participants will be asked to use a gel pillow with a cooling surface the night before the day of surgery.

If there is a comparison group: Researchers will compare patients' control group to see if there is any difference in sleep quality and comfort levels.

DETAILED DESCRIPTION:
Randomization method will be used to determine the groups. Randomization of the patients was done using the 'Random Allocation Software 2.0' program and they are allocated into 2 groups: 1) the control group and 2) the intervenion group.

1. The Control Group: The patients in this group will be visited by the researcher in their rooms on the morning before the surgery. Patients will be informed that they will be visited again in the evening of the day before the surgery and that they will be given a pillow to use while sleeping at night. They will receive no other interventions.Patients will be visited again on the morning of the surgery day.The Richard Campbell Sleep Scale was used to evaluate the nighttime sleep quality of the patients;General Comfort Scale to evaluate comfort levels.
2. The Intervenion Group: The patients in this group will be visited by the researcher in their rooms on the morning before the surgery. Patients will be informed that they will be visited again in the evening of the day before the surgery and that they will be given a pillow to use while sleeping at night. Patients who are visited in their rooms on the evening of the day before the surgery will be given a gel pillow with a cooling surface feature for night use. If patients stop using pillows at night, they will be asked to inform the investigator when they come to their room in the morning.Patients will be visited again on the morning of the surgery day.The Richard Campbell Sleep Scale was used to evaluate the nighttime sleep quality of the patients;General Comfort Scale to evaluate comfort levels.

ELIGIBILITY:
Inclusion Criteria:

To research;

* Planned elective surgery
* Those who will undergo cancer surgery related to the gastrointestinal system
* No diagnosis of sleep disorder
* No sensory, cognitive or mental disability
* Using pillows while sleeping
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* Emergency surgical intervention will be performed
* In contact isolation
* The one who has given up using a gel pillow for sleep at night
* Diagnosis of diseases related to the endocrine system (such as diabetes, obesity)
* Using hormone replacement medication
* Patients using anti-depressant medication were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Sleep quality level | 12 mounth
  Sleep quality of the patietns will be evaluated with Richards Campbell Sleep Scale. Each item in the scale is evaluated on a chart between 0 and 100 using the visual analog scale technique. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. The high score of the scale indicates that the sleep quality of the patients is high.

SECONDARY OUTCOMES:
Comfort level | 12 mounth
  Comfort level of the patietns will be evalueated with General Comfort Scale. The lowest total score that can be obtained from the scale is 48, and the highest total score is 192. The average value is determined by dividing the total score obtained by the number of scale items, and the result is indicated in the 1-4 distribution. Low comfort is expressed by one point, high comfort by four points.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Principal Investigator — Trakya University; Esra Çevik, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No